CLINICAL TRIAL: NCT03314753
Title: FIRE AND ICE Re-Ablations: Retrospective Data Collection on Re-ablations Performed Within the FIRE AND ICE Trial
Brief Title: FIRE AND ICE Re-Ablations (Retrospective Data Collection)
Acronym: Re-Do
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17038
Record Dates: First submitted 2017-09-25; First posted 2017-10-19 (Actual); Results first posted 2019-09-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cryoballoon Arm from FIRE AND ICE Trial: No new/additional patients will be enrolled within this project. Only retrospective data will be collected on performed re-ablation procedures within the FIRE AND ICE Trial.
  The FIRE AND ICE Trial collected data to compare efficacy and safety of isolation of the pulmonary veins (PV) using a Cryoballoon catheter versus (Cryoballoon Arm) a radiofrequency ablation (RF Arm) with a ThermoCool catheter in patients with drug refractory symptomatic paroxysmal atrial fibrillation (AF).
  Products Used within the FIRE AND ICE Trial: Arctic Front® & Arctic Front Advance® Cardiac CryoAblation Catheter System.
  The purpose of this retrospective data collection on re-ablations performed in both treatment arms (Cryo arm and Radiofrequency arm) of the FIRE AND ICE Trial.
  Interventions: Other: No interventions - retrospective data collection
- Radiofrequency Arm from FIRE AND ICE Trial: No new/additional patients will be enrolled within this project. Only retrospective data will be collected on performed re-ablation procedures within the FIRE AND ICE Trial.
  The FIRE AND ICE Trial collected data to compare efficacy and safety of isolation of the pulmonary veins (PV) using a Cryoballoon catheter versus (Cryoballoon Arm) a radiofrequency ablation (RF Arm) with a ThermoCool catheter in patients with drug refractory symptomatic paroxysmal atrial fibrillation (AF).
  Products Used within the FIRE AND ICE Trial: NaviStar® ThermoCool® Ablation Catheter (Radiofrequency Arm; Manufacturer Biosense Webster, Inc.).
  The purpose of this retrospective data collection on re-ablations performed in both treatment arms (Cryo arm and Radiofrequency arm) of the FIRE AND ICE Trial.
  Interventions: Other: No interventions - retrospective data collection

INTERVENTIONS:
Other: No interventions - retrospective data collection — No new patients will be enrolled within this project; only retrospective data will be collected on performed re-ablations within the FIRE AND ICE Trial

SUMMARY:
Retrospective data collection on re-ablations performed within the FIRE AND ICE Trial.

DETAILED DESCRIPTION:
The purpose of this retrospective data collection on re-ablations performed in both treatment arms (Cryo arm and Radiofrequency arm) of the FIRE AND ICE Trial is to gain insight into re-occurrence of atrial arrhythmias resulting in a re-ablation after a performed index ablation procedure. Data to be collected from subject charts include pulmonary vein anatomy, documented atrial arrhythmias prior to re-ablation, pulmonary vein reconnection, pulmonary vein ablation lesion gaps and gap location, ablation lesions performed during the re-ablation, procedure parameters of the RF or cryo catheter utilized during the re-ablation, and success of re-ablations performed.

ELIGIBILITY:
N/A - no new patients will be enrolled within this project.

Inclusion Criteria for the FIRE AND ICE Trial included:

* Symptomatic paroxysmal atrial fibrillation (PAF) with at least two episodes and at least one episode documented (30 seconds episode length, documented by electrocardiogram (ECG) within last 12 months
* Documented treatment failure for effectiveness of at least one anti-arrythmic drug (AAD Type I or III, including Beta-Blocker and AAD intolerance)
* 18 to 75 years of age
* Patients who are mentally and linguistically able to understand the aim of the trial and to show sufficient compliance in following the trial protocol
* Patient is able to verbally acknowledge and understand the associated risks, benefits, and treatment alternatives to therapeutic options of this trial: cryoballoon ablation system or standard radiofrequency (RF) ablation technique.

The exclusion criteria were grouped as follows in the FIRE AND ICE Trial:

* General exclusion criteria
* Exclusion criteria related to the cardiac condition
* Exclusion criteria based on laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The FIRE AND ICE Trial collected data to compare efficacy and safety of isolation of the pulmonary veins (PV) using a Cryoballoon catheter versus a radiofrequency ablation with a ThermoCool catheter in patients with drug refractory symptomatic paroxysmal atrial fibrillation (PAF).
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Nemocnice Na Homolce Praha, Prague, Czechia
- Clinique Pasteur Toulouse, Toulouse, France
- Germany (5):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Cardioangiologisches Centrum Bethanien CCB, Frankfurt am Main
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Herz-Zentrum Bodensee, Konstanz
- Isala Klinieken Zwolle, Zwolle, Netherlands
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico San Carlos Madrid, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario Valencia, Valencia
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuck KH, Albenque JP, Chun KJ, Furnkranz A, Busch M, Elvan A, Schluter M, Braegelmann KM, Kueffer FJ, Hemingway L, Arentz T, Tondo C, Brugada J; FIRE AND ICE Investigators. Repeat Ablation for Atrial Fibrillation Recurrence Post Cryoballoon or Radiofrequency Ablation in the FIRE AND ICE Trial. Circ Arrhythm Electrophysiol. 2019 May 22;12(6):e007247. doi: 10.1161/CIRCEP.119.007247. PMID 31693319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 110 patients reported a re-ablation in the original FIRE AND ICE Trial. Of those 110, 89 consented for the FIRE AND ICE Re-Ablation study. All data available in retrospective chart review from the 89 subjects were included in analyses. No patient data was excluded.
  The first re-ablation for each patient was included in the analysis.
Groups:
- Radiofrequency Arm From FIRE AND ICE Trial: No new/additional patients will be enrolled within this project. Only retrospective data will be collected on performed re-ablation procedures within the FIRE AND ICE Trial.
  The FIRE AND ICE Trial collected data to compare efficacy and safety of isolation of the pulmonary veins (PV) using a Cryoballoon catheter versus (Cryoballoon Arm) a radiofrequency ablation (RF Arm) with a ThermoCool catheter in patients with drug refractory symptomatic paroxysmal atrial fibrillation (AF).
  Products Used within the FIRE AND ICE Trial: NaviStar® ThermoCool® Ablation Catheter (Radiofrequency Arm; Manufacturer Biosense Webster, Inc.).
  The purpose of this retrospective data collection on re-ablations performed in both treatment arms (Cryo arm and Radiofrequency arm) of the FIRE AND ICE Trial.
  No interventions - retrospective data collection: No new patients will be enrolled within this project; only retrospective data will be collected on performed re-ablations within the FIRE AND ICE Trial
- Cryoballoon Arm From FIRE AND ICE Trial: No new/additional patients will be enrolled within this project. Only retrospective data will be collected on performed re-ablation procedures within the FIRE AND ICE Trial.
  The FIRE AND ICE Trial collected data to compare efficacy and safety of isolation of the pulmonary veins (PV) using a Cryoballoon catheter versus (Cryoballoon Arm) a radiofrequency ablation (RF Arm) with a ThermoCool catheter in patients with drug refractory symptomatic paroxysmal atrial fibrillation (AF).
  Products Used within the FIRE AND ICE Trial: Arctic Front® & Arctic Front Advance® Cardiac CryoAblation Catheter System.
  The purpose of this retrospective data collection on re-ablations performed in both treatment arms (Cryo arm and Radiofrequency arm) of the FIRE AND ICE Trial.
  No interventions - retrospective data collection: No new patients will be enrolled within this project; only retrospective data will be collected on performed re-ablations within the FIRE AND ICE Trial
Period: Overall Study
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Started | 53 | 36
Completed | 53 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial | Total
Number analyzed (Participants) | 53 | 36 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (10) | 62 (11) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 33 | 15 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 5 | 1 | 6
  Czechia | 3 | 0 | 3
  France | 1 | 1 | 2
  Switzerland | 2 | 5 | 7
  Germany | 34 | 25 | 59
  Spain | 8 | 4 | 12
Diagnosed with paroxysmal atrial fibrillation (PAF) [year] [Mean (Standard Deviation); unit: years] | 6.1 (6.5) | 5.5 (4.5) | 5.9 (5.7)
BodyMassIndex (BMI) [kg/m^2] [Mean (Standard Deviation); unit: kg/m^2] | 27 (4) | 28 (5) | 28 (4)
Height [cm] [Mean (Standard Deviation); unit: cm] | 176 (10) | 170 (9) | 173 (10)
Weight [kg] [Mean (Standard Deviation); unit: kg] | 85 (16) | 81 (15) | 83 (15)
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) Functional Classification provides a way of classifying the extent of heart failure.
  NYHA I - No limiation of phyiscal activity. NYHA II - Slight limiation of phyiscial activity. NYHA III - Marked limiation of physical activity. NYHA IV - Unable to carry on any physical activity without discomfort. Within FIRE AND ICE Re-Do the majorty of patients 69% does not have heart failure signs. If any signs of heart failure documented in the baseline, then only mild forms. No heart failure patients (NYHA III or IV) were seen/enrolled in FIRE AND ICE Re-Do.
  Participants
    Patient does not have heart failure | 39 | 22 | 61
    NYHA Class I | 3 | 4 | 7
    NYHA Class II | 11 | 10 | 21
    NYHA Class not available | 0 | 0 | 0
Left Atrial Diameter (LAD) [mm] [Mean (Standard Deviation); unit: mm] — Left Atrial Diameter was measured within the trial. An anteroposterior left atrial diameter of more than 55 mm as measured by trans-thoracic echocardiography is an exclusion criteria within the inital FIRE AND ICE Trial (outcome of ablation in patients with significant atrial dilation > 55 mm is lacking data but is seen as possible predictor for pulmonary vein isolation failure/atrial fibrillation recurrence).
  mm | 41.6 (5.7) | 39.4 (7.9) | 40.6 (6.8)
Left Ventricular Ejection Fraction (LVEF) [%] [Mean (Standard Deviation); unit: %] — The ejection fraction (EF) is a measurement, expressed as percentage, of how much blood the left ventricle pumps out with each contraction, e.g. an ejection fraction of 60% means that 60% of the total amount of blood in the left ventricle is pushed out with each heartbeat.
  Therefore the ejection fraction is an indcation of how well the heart is pumping and may be an evidence of heart failure (under 40%) or cardiomyopathy.
  % | 62 (7) | 62 (7) | 62 (7)
Left Ventricular End Diastolic Diameter (LVEDD) [mm] [Mean (Standard Deviation); unit: mm] | 51 (4) | 51 (5) | 51 (5)
Left Atrium (LA) Volume [mL] [Mean (Standard Deviation); unit: mL] | 73 (35) | 62 (41) | 69 (36)
Prior Direct Current Cardioversion (DCCV) [Number; unit: participants] | 15 | 8 | 23
History of Atrial Flutter [Number; unit: participants] | 11 | 6 | 17
Prior Stroke [Number; unit: participants] | 2 | 2 | 4
Coronary Artery Disease (CAD) [Number; unit: participants] | 3 | 1 | 4
Prior Myocardial Infarction (MI) [Number; unit: participants] | 1 | 0 | 1
Aortic Valve Stenosis [Number; unit: participants] | 0 | 0 | 0
Peripheral Artery Disease [Number; unit: participants] | 0 | 0 | 0
Hyperlipidemia [Number; unit: participants] | 13 | 12 | 25
Diabetes Type I or II [Number; unit: participants] | 5 | 4 | 9
Hypertension [Number; unit: participants] | 32 | 22 | 54
Prior Coronary Artery Bypass Graft (CABG) [Number; unit: participants] | 2 | 0 | 2
Prior Percutaneous Coronary Intervention (PCI) [Number; unit: participants] | 2 | 0 | 2
Antiarrhythmic Druc (AAD) at discharge [Number; unit: participants] | 18 | 14 | 32
HATCH Score [Mean (Standard Deviation); unit: units on a scale] — The HATCH score stratifies patients with paroxysmal atrial fibrillation according to their risk for progression of sustained atrial fibrillation within 1-year.
  The HATCH score is an ordinal scale ranging from 0 to 7 points and is calculated based on the following formula: 1x (Hypertension) + 1 x (Age >75years) + 2 x (Transient Ischemic Attack or Stroke) + 1x (Chronic Obstructive Pulmonary Disease) + 2x (Heart Failure).
  Higher HATCH score is seen in literature as increased risk for progression of sustained atrial fibrillation.
  units on a scale | 1.2 (1.1) | 1.5 (1.2) | 1.3 (1.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHG] | 134 (24) | 133 (22) | 134 (23)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHG] | 79 (13) | 76 (11) | 78 (12)
Glomerular Filtration Rate (GFR) [Mean (Standard Deviation); unit: mL/min/m2] | 75 (16) | 77 (19) | 76 (17)
CHA2DS2-VASc [Mean (Standard Deviation); unit: units on a scale] — CHA2DS2-VASc Score for Atrial Fibrillation Stroke Risk.
  Score is between 0 and 9 points:
  1 point - Congestive Heart Failure
  1 point - Hypertension 2 point - Age > 75 years
  1. point - Diabetes mellitus
  2. point - Stroke / Transient Ischemic Attach / Thromboembolic Event
  1 point - Vascular Disease (prior myocardial infarction, peripheral artery disease, or aortic plaque)
  1 point - Age 65 to 74 years
  1 point - Sex category (i.e. female sex)
  A high score is the same as a higher stroke risk, and a low score means the lower stroke risk.
  units on a scale | 1.8 (1.3) | 2.3 (1.3) | 2.0 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Documented Atrial Arrhythmias Prior to Re-ablation
Description: Number of documented atrial arrhythmias as assessed by ECG prior to the re-ablation
Time Frame: At time of re-ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
Participants
  Paroxysmal Atrial Fibrillation (PAF) | 36 | 25
  Persistent Atrial Fibrillation | 7 | 5
  Atrial Tachycardia (AT)/Atrial Flutter (AFL) | 6 | 5
  Atrial Fibrillation/Supraventricular Tachycardia | 3 | 0
  Other | 1 | 1

2. Primary Outcome: Number of Reconnected Pulmonary Veins as Documented in the Cath Lab / Imaging at the Time of Re-ablation Procedure
Description: Number of reconnected pulmonary veins as documented in cath lab / imaging
Time Frame: At time of re-ablation
Measure: Mean (Standard Deviation); unit: Reconnected Pulmonary Veins
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
Reconnected Pulmonary Veins | 2.1 (1.4) | 1.4 (1.1)

3. Primary Outcome: Number of Gaps and Location of Gaps Present in Pulmonary Vein Ablation Lesions Per Participant
Description: Number of gaps and location of gaps present in pulmonary vein ablation lesions as seen in the cath lab / imaging
Time Frame: At time of re-ablation
Population: Data were not collected; no standard documention and therfore not available in the reviewed medical files in the required detail
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number of Pulmonary Veins Ablation - Ablation Lesion Sets Created During Re-ablation Procedure
Description: Description of all ablation lesion sets created during re-ablation procedure
Time Frame: At time of re-ablation
Population: The number of lesion sets for each patient was counted for this objective. If a patient had multiple pulmonary veins ablated during the re-ablation procedure, each pulmonary vein was counted as a lesion set towards the patients total count.
Measure: Mean (Standard Deviation); unit: Pulmonary Veins ablated
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
Pulmonary Veins ablated | 2.4 (1.4) | 1.8 (1.4)

5. Primary Outcome: Percentage of Participants With Acute Procedural Success of Re-ablation Procedure
Description: Summarize acute procedural success of re-ablation procedure per treatment arm
Time Frame: At time of re-ablation
Population: A patient was defined as an acute success if all ablation attempts within the re-ablation procedure were reported as successful. Pulmonary Vein Isolation (PVI) was assessed minimally via documented entrance block, and where assessable exit block (electrical signal detection).
Measure: Number; unit: percentage of patients with acute succes
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
percentage of patients with acute succes | 90.4 | 93.9

6. Primary Outcome: Re-ablation Procedure Times as Measured in the Cath Lab
Description: Re-ablation procedure times as measured in the cath lab
Time Frame: At time of re-ablation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
minutes | 122 (53) | 103 (33)

7. Primary Outcome: Number of Hospital Days for Re-ablation Procedure Form Admission to Discharge
Description: Number of hospital days for re-ablation procedure form admission to discharge
Time Frame: From Date of Hospital admission until the date of hospital discharge up to 36 month FU period
Measure: Mean (Standard Deviation); unit: nights
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
nights | 2.6 (2.1) | 2.5 (2.7)

8. Primary Outcome: Number of Participants With Anti-arrhythmic Drug Use at Time of Discharge From the Re-ablation Procedure
Description: Anti-arrhythmic drug use at time of discharge from the re-ablation procedure via medical log on AADs
Time Frame: Date of hospital discharge, assessed during the 36 month FU period
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
Participants | 30 | 19

9. Primary Outcome: Number of Participatns With Adenosine Testing
Description: Number of participants with adenosine testing
Time Frame: At time of re-ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
Number analyzed (Participants) | 53 | 36
Participants | 10 | 4

ADVERSE EVENTS:
Time Frame: Within this retrospective data collection, no additional or new safety data was collected. Safety reporting on all events was already performed as part of the original FIRE AND ICE Trial.
Description: Not applicable. Safety reporting on all events was already performed as part of the original FIRE AND ICE Trial.
Arm/Group | Radiofrequency Arm From FIRE AND ICE Trial | Cryoballoon Arm From FIRE AND ICE Trial
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications from this retrospective data collection are regulated separately in the publication plan, which was reviewed and approved by the Publication Committee.

Medical Centers / Investigators may publish the results of work performed under the applicable site agreement. Any such publication shall be at a time determined by Medtronic and shall be provided to Medtronic for review at least 60 days prior to submission or presentation.

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/53/NCT03314753/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT03314753/SAP_001.pdf